CLINICAL TRIAL: NCT06323317
Title: The Feasibility and Triability of a Prehabilitation Program for Mild to Moderately Frail Patients Undergoing Cardiac Surgeries/Procedures
Brief Title: A Prehabilitation Program for Frail Patients Undergoing Cardiac Surgeries/Procedures
Acronym: PREHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW 21-405
Record Dates: First submitted 2024-03-03; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Bypass Grafting; Heart Valve Replacement; Transcatheter Aortic Valve Implantation; Frailty
Keywords: prehabilitation; home-based exercise; centre-based exercise; coronary artery bypass grafting; valve replacement; valve repair; transcatheter aortic valve implantation; cardiac patients
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The post-intervention data collector (research assistant) will be blinded to the group allocation to avoid performance and detection biases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frailty-Specific Prehabilitation Program (Experimental): Participants in the frailty-specific prehabilitation program (intervention group) will participate in a comprehensive prehabilitation programme comprising the following components: 1) structured preoperative education; 2) nutritional optimization; 3) stress management; and 4) exercise training. These four components are recommended by the international association as core elements of prehabilitation to optimize cardiac patients' physical and psychological capacity to withstand the challenges of cardiac surgical procedures. The prehabilitation will last for at least 4 weeks, and it will continue throughout the preoperative period.
  Interventions: Behavioral: Multi-component exercise programme; Behavioral: Structured preoperative education; Behavioral: Nutritional optimization; Behavioral: Stress management
- Routine Preoperative Care (Placebo Comparator): Participants in the control group will receive routine preoperative care provided by the clinical team, which includes unstructured patient education on the surgeries/procedures, and a brief session on the use of an incentive spirometer, breathing, and coughing exercise. Other perioperative care procedures will be implemented according to the existing clinical protocols.
  Interventions: Other: Attention Placebo

INTERVENTIONS:
Behavioral: Multi-component exercise programme — Each exercise session will start with a warm-up, followed by core exercise training and ending with a cool-down period. A series of flexibility training and stretching exercises will be performed during the warm-up and cool-down phases (10 minutes in total). The core exercise session will comprise aerobic (10 minutes), resistance (20 minutes), and balance (20 minutes) training, where resistance and balance exercises constitute the major components, as they are particularly effective in strengthening functional capacity, muscle strength, and balance function for mobility in frail patients.
  Arms: Frailty-Specific Prehabilitation Program
Other: Attention Placebo — The control group will receive routine preoperative care provided by the clinical team, which includes unstructured patient education on the surgeries/procedures, and a brief session on the use of an incentive spirometer, breathing, and coughing exercise. Other perioperative care procedures will be implemented according to the existing clinical protocols.
  Arms: Routine Preoperative Care
Behavioral: Structured preoperative education — The prehabilitation programme will begin with a 60-minute (group- or individual-based) structured education session at the centre. The content will cover frailty, its impacts on postoperative recovery, cardiovascular and overall health, and functional well-being. The importance of nutrition and exercise on their recovery potential and postoperative functional capacity will be elaborated. Their commitment to intervention engagement will be highlighted as the key to success. This session will also cover the principles of exercise, its progression, and exercise safety.
  Arms: Frailty-Specific Prehabilitation Program
Behavioral: Nutritional optimization — The Malnutrition Universal Screening Tool (MUST) will be used for a nutritional screening to determine the risk of malnutrition (low, medium, or high). The nurse will evaluate the dietary patterns of each participant, and provide tailored nutritional advice on daily protein intake according to a protein supplementation protocol. The participants and their caregivers will be provided with plenty of suggestions for high-quality protein foods according to patients' preferences. The nurse will follow-up with the participants to identify any barriers they encountered in real-world settings when they attend the exercise sessions. She will reinforce the advice and provide suggestions to overcome barriers according to the preference and lifestyle of the participants.
  Arms: Frailty-Specific Prehabilitation Program
Behavioral: Stress management — Relaxation techniques to reduce tense arousal, including guide imagery and breathing techniques, will be taught. Guided imagery makes use of attention-focus to target mental arousal, whereas deep and diaphragmatic breathing is a fundamental relaxation method for various stress relieving techniques. Both techniques are designed to reduce sympathetic arousal, which is particularly beneficial to cardiac patients. Participants will be encouraged to self-practice on a daily basis, and a sound track will be provided to guide their practice.
  Arms: Frailty-Specific Prehabilitation Program

SUMMARY:
The purpose of this study is to develop and evaluate a frailty-specific prehabilitation program for patients awaiting cardiac surgeries/procedures. The program aims to improve functional capacity, frailty level, cardiac-related physical functioning, health-related quality of life (HRQoL), psychological distress, major adverse cardiovascular and cerebral events (MACCE), hospital length of stay, and readmission rates.

Cardiovascular disease is a leading cause of disability and morbidity globally, particularly in older adults. Frailty, a geriatric syndrome commonly seen in cardiac patients, complicates their perioperative care and leads to worse outcomes.

Prehabilitation, which optimizes patients' physiological and functional capacities before surgery, has shown promise in general cardiac patients but requires a more comprehensive approach for frail individuals. This randomized controlled trial will recruit 50 Chinese adults awaiting elective cardiac surgeries/procedures in Hong Kong. Participants will be randomly assigned to either the intervention group, receiving a comprehensive prehabilitation program, or the control group, receiving routine preoperative care. Assessments will be conducted at baseline and at three postoperative time points.

The findings will contribute to our understanding of the impact of frailty on postoperative outcomes and help develop strategies to improve patient care. Ultimately, this study aims to reduce healthcare burdens associated with cardiac disease-related morbidity and disability.

DETAILED DESCRIPTION:
Cardiovascular disease is a major cause of disability and morbidity worldwide. With advances in medical technology and care, patients with cardiovascular disease often live to an advanced age. In the older cohort, conditions particularly associated with age-related atherosclerosis and calcification dominate, such as coronary artery disease and valvular heart disease. Surgical interventions remain the treatment-of-choice for patients with advanced cardiac conditions. However, this vulnerable cohort is still afflicted by a higher risk of mortality, postoperative complications, and longer hospital stays, particularly those with frailty.

Frailty is a clinical condition characterized by reduced reserve capacity and excessive vulnerability to increased risk of adverse health outcomes when exposed to stressors. Its prevalence increases in the population with cardiovascular disease and is a significant prognostic indicator for predicting postoperative outcomes in cardiac patients. The best strategy to minimize the prognostic impacts of frailty on cardiac patients should be intervened at the preoperative stage, which may be achieved through prehabilitation.

Prehabilitation refers to preoperative interventions designed to optimize patients' physical and psychological readiness for surgery. The international guidelines of the Enhanced Recovery After Surgery Society (ERAS) suggest the prehabilitation for cardiac surgical patients should be exercise-based, supplemented with education, dietary modification, and psychological support. These components can prepare patients to withstand stressful events during surgery through reducing sympathetic over-activity and improving their physiological and functional capacities.

Accumulating evidence indicates the effectiveness of prehabilitation for general cardiac patients through respiratory muscle and aerobic training; however, few studies have investigated those with frailty, who are in greater need. Among the limited trial that particularly focus on frail patients, encouraging findings have been reported that preliminarily indicate their efficacy and safety profile. There are also some ongoing trials testing prehabilitation for frail cardiac patients registered in trial registries.

Despite the promising results, there are several major knowledge gaps in the studies of prehabilitation for frail cardiac patients. First, most of these trials are testing a single frailty-reversing strategy, either nutritional or exercise interventions, which are less comprehensive to address the urgent needs of surgical patients. Second, the protocols of those exercise programs are mainly aerobic-focused, deviating from the principles of exercise prescription suggested for frailty management. Third, all completed and ongoing trials are center-based using gymnasium equipment, which has several limitations that jeopardize the feasibility, availability, and effectiveness of the programs.

To conclude, more comprehensive and accessible prehabilitation programs are needed for frail cardiac patients to address their complex needs and improve their surgical outcomes. A hybrid approach, using eHealth to supplement in-person patient support, could offer a more practical and feasible solution. Further research is required to develop and evaluate such programs and to fill the knowledge gaps in prehabilitation for frail cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed schedule for elective CABG, valve repair/replacement, or combined CABG and valve repair/replacement, or TAVI
2. Mild to moderate frailty at the time of recruitment, indicated by a Clinical Frailty Scale score between 4 and 6
3. At least 5 weeks of procedural waiting time
4. Physically fit for prehabilitation according to the surgeon/cardiologist's endorsement on a risk-assessment checklist
5. Living with family
6. Using an electronic device with internet access (patient/family).

Exclusion Criteria:

1. Impaired cognition (Abbreviated Mental Test score ≤6) or communication
2. With physical limitations to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  It is used to assess functional capacity. A brief performance-based assessment consisting of 3 timed-tasks, namely standing balance, walking speed, and chair stand tests. The timed results will be rescaled to obtain a score ranging from 0 to 12, with higher scores indicating better functional status.
Weakness/ Grip Strength (Fried Phenotype Frailty Assessment) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  (For Outcome measures 2 to 6): Fried Phenotype Frailty Assessment consists of five domains (Outcome 2 to Outcome 6). If the aggregated score is (3-5), the subject is classified as being frail. Fried Phenotype Frailty Assessment is a valid, reliable, and commonly used tool for assessing frailty.
  Weakness is measured by the maximal grip strength (kilograms) in the dominant hand (3 measures averaged), using a hand-held dynamometer. This criterion is met if grip strength is measured at the lowest 20% at baseline, adjusted for gender and body mass index.
Slowness (Fried Phenotype Frailty Assessment) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  Slowness is measured by using the 5-meter walking test. This criterion is met for the slowest 20% of the population at baseline, based on the time to walk 5 metres, adjusting for gender and standing height.
Low Physical Activity (Fried Phenotype Frailty Assessment) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  The Minnesota Leisure Time Activities Questionnaire is used to measure physical activities in the prior 2 weeks, plus frequency and duration. Physical function was measured by asking about difficulty with 15 tasks of daily life, including mobility, upper extremity, instrumental activities of daily living (IADL). A weighted score of kilocalories expended per week was calculated at baseline based on each participant's report. This criterion is met if the kilcalories expenditure is below the cut-off values as described by Fried and colleagues (men 383 kcal/week, women 270 kcal/week).
Self-reported Exhaustion (Fried Phenotype Frailty Assessment) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  Exhaustion is measured by using two items from the Center for Epidemiological Studies Depression scale: "How often did you feel that everything you did was an effort?" and "How often did you feel that you could not get going?" This criterion was met when participants answered: "always or most of the times" to at least one of the two questions.
Unintentional Weight Loss (Fried Phenotype Frailty Assessment) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  Weight loss is measured by calculating if the subject has lost at least 5 percent of previous year' body weight unintentionally (i.e. not due to dieting or exercise). This criterion is met if unintentional weight loss ≥ 5 percent.
The Seattle Angina Questionnaire (SAQ) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  It is used to measure cardiac-related functional status. It has 19 items in 5 subscales: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. It is scored on a 1-5 or 6 sequentially coded scale, and subscale scores are transformed to a scale of 0-100, with higher scores indicating higher levels of functioning and fewer limitations. The Chinese version has been shown to be reliable, valid, and sensitive to clinical change.
The MacNew Heart Disease Health-Related Quality of Life Questionnaire | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  The MacNew will be used to measure cardiac-specific HRQoL. It has 27 items scored on a 1-7 Likert scale, ranging from "all of the time" to "some of the time", with higher score representing better HRQoL. A global score is then calculated by averaging the item scored (from 1-7), with higher scores also representing better HRQoL. MacNew has good internal consistency, test-retest reliability, and concurrent and discriminant validity.

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  It is used to measure anxiety and depression. It has 14 items in two subscales scored on a 4-point Likert scale, with higher scores indicating a more intensive anxious and depressed mood. It has good internal consistency and concurrent and criterion validity.
Biomarkers-Serum albumin | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  Serum albumin count (mg/dL) will be collected according to standard laboratory guidelines in the clinical setting.
Biomarkers- C-reactive protein | At baseline (T0), one-day before surgery (T1), postoperative 1 month (T2), and postoperative 3 months (T3)
  C-reactive protein count (mg/L) will be collected according to standard laboratory guidelines in the clinical setting.
Major adverse cardiac and cerebrovascular events (MACCE) | Monitored from Day 0 to 3 months postoperative through record review
  Document through record review
Hospital Length of stay | Monitored from Day 0 to 3 months postoperative through record review
  Document through record review
Hospital Readmissions | Monitored from Day 0 to 3 months postoperative through record review
  Document through record review

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Dr, Principal Investigator — The University of Hong Kong, School of Nursing
Locations (1):
- Polly Wai Chi, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No